CLINICAL TRIAL: NCT05076643
Title: Biomarkers, Traditional Chinese Medicine Body Constitution, Dietary Pattern and Psychological Factors in Predicting Depression Among University Students in UTAR, Malaysia
Brief Title: Biomarkers, TCM Body Constitution, Dietary Pattern and Psychological Factors in Predicting Depression
Status: Recruiting | Type: Observational
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Foo Chai Nien, Assistant Professor, Universiti Tunku Abdul Rahman
Other Study IDs: IPSR/RMC/UTARRF/2019-C2/F01
Record Dates: First submitted 2021-09-30; First posted 2021-10-13 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- University students: University students in Universiti Tunku Abdul Rahman Sungai Long Campus

SUMMARY:
This study aims to determine the predictors of depression among university students in Universiti Tunku Abdul Rahman (UTAR) Sungai Long Campus.

DETAILED DESCRIPTION:
University students are a high at risk group for development of depression. Identifying the determinants of depression could help in the diagnosis and treatment of this disorder. This study will incorporate questionnaire and blood sample data collection procedures on 397 subjects. Written consent will be obtained from the subjects. Eligible subjects will be given self-administered questionnaires which include Patient health questionnaire (PHQ-9), Constitution in Chinese medicine questionnaire (CCMQ), Dysfunctional Attitude Scale (DAS), Depression Anxiety Stress Scales (DASS-21) - stress and anxiety subscales, Perceived stress scale-10 (PSS-10), Rosenberg self-esteem scale (RSES), and Food frequency questionnaire (FFQ). Once the subjects completed the questionnaires, blood samples will be collected from them by a trained phlebotomist. In addition, 10 most high at risk of depression subjects (with PHQ-9 scores 10 and above) and 10 healthy subjects (with PHQ-9 scores lower than 10) will be selected randomly for protein expression to further identify the proteins that significantly expressed among them.

ELIGIBILITY:
Inclusion Criteria:

* Malaysian citizen
* Able to read and communicate in English

Exclusion Criteria:

* Special education disability (deaf and blind)
* Physical support
* History of infectious diseases

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: University students
Sampling Method: Probability Sample
Enrollment: 397 (Estimated)
Dates: Start 2022-03-17 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Genetic, TCM body constitution, psychological factors and dietary pattern are significant predictors for depression among university students. | Baseline
  Univariate and multivariate logistic regression will be performed.

SECONDARY OUTCOMES:
Prevalence of depression among university students. | Baseline
  Patient Health Questionnaire (PHQ-9):
  Non depressed = 0 - 9; Depressed = 10 - 27
Protein significantly expressed between depressed and non-depressed students. | Baseline
  Liquid chromatography-mass spectrometry (LC-MS) will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Chai Nien Foo, Principal Investigator — Universiti Tunku Abdul Rahman
Locations (1):
- Universiti Tunku Abdul Rahman, Kajang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No